CLINICAL TRIAL: NCT06295029
Title: Dose Optimization and Personalized Medication Software Research of BCL-2 Inhibitor Based on Machine Learning Combined With Genomics in Patients With Acute Myeloid Leukemia
Brief Title: Personalized Medication Software for BCL-2 Inhibitor in AML Patients Using Machine Learning and Genomics
Status: Not yet recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: CPA-Z05-ZC-2023-002
Record Dates: First submitted 2024-02-26; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Venetoclax; Machine Learning; genomics; Dose Prediction; Personalized medicine
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two ml of peripheral blood samples from patients were placed in Ethylenediaminetetraacetic acid(EDTA) tubes,DeoxyriboNucleic Acid(DNA) was extracted and cryopreserved for use in the determination of relevant SNPs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe neutropenia caused by venetoclax,a B-cell lymphoma-2(BCL-2) inhibitor, is the main cause of venetoclax tapering, drug discontinuation, and treatment delay. This study combines machine learning and genomics, hoping to develop models to predict venetoclax dose in Acute myeloid leukemia(AML) patients and compare the efficacy and safety differences of model-guided individualized medication regimen with current conventional regimen. According to the demographic information, the drug information, the drug concentration of the target patients, the laboratory examination, the single nucleotide polymorphism(SNP) information and the adverse reactions of the AML patients, and the model was constructed through machine learning.

DETAILED DESCRIPTION:
Introduction:The successful development of venetoclax offers new hope for AML patients not eligible for strong induction chemotherapy. However, there are some clinical problems, such as severe neutropenia is the main reason for treatment delay and discontinuation of patients. The Asian population has higher drug exposure than the non-Asian population, and the blood concentration of venetoclax varies greatly individually, and the blood drug concentration is associated with efficacy and adverse effects. We urgently need an individualized study of venetoclax for Chinese AML patients to reduce the incidence of adverse events while ensuring efficacy.

Objective：Construction of a venetoclax dose prediction model for AML patients based on machine learning combined genomics;

Methods：1.Venetoclax plasma concentration determination;determination of SNPs of related genes in patient blood cells; 2.venetoclax dose prediction model for AML patients based on machine learning techniques combined with genomics Collect the clinical data and establish a database Mining variables to explore the factors affecting the dosage of venetoclax Building a predictive model based on a machine-learning algorithm Model performance was evaluated, and the optimal model was selected Interpretation and optimization of the model

The AML patients were conditionally screened by the study physician involved in the project department to assess their enrollment. Communicate fully with the patients and their family members who meet the enrollment criteria, obtain the patient's informed consent, and sign the informed consent form. After enrollment, patient clinical data were recorded. Evaluation according to the efficacy and safety evaluation criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, regardless of gender;
2. Diagnosed as an AML patient according to the Diagnosis and Treatment Guidelines for Adult Acute Myeloid Leukemia (Non Acute Promyelocytic Leukemia) in China (2021 Edition) and receiving treatment with venetoclax;
3. Before receiving venetoclax treatment, absolute neutrophil count (ANC) ≥ 1.0 ×10 ^9/L, white blood cell count (WBC) ≥ 2.0 ×10 ^9/L, platelet count (PLT) ≥ 50 ×10 ^9/L, and hemoglobin (HB) ≥ 90g /L;
4. Before receiving venetoclax treatment, liver and kidney function were normal (aspartate aminotransferase ≤ 3 times the upper limit of normal (ULN), alanine aminotransferase ≤ 3.0 x ULN, bilirubin ≤ 1.5 x ULN, urea nitrogen:3.2-7.1 mmol/L, glomerular filtration rate (eGFR) ≥ 60ml/min;
5. Sign an informed consent form.

Exclusion Criteria:

1. Age<18 years old;
2. Non AML patients;
3. Patients who plan to use a treatment regimen without venetoclax;
4. Patients with poor medication adherence;
5. Liver and kidney function damage before medication;
6. Before medication, ANC<1.0 x 10 ^9/L or WBC<2.0 x 10 ^9/L or PLT<50 x 10 ^9/L or HB<90g /L;
7. Pregnant and lactating women;
8. Cases deemed unsuitable for inclusion by researchers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to include 200 patients with AML who were treated with venetoclax. A database of venetoclax medication for AML patients will be constructed based on demographic information, medication information, laboratory test information, blood drug concentration, SNPs, and drug-related adverse reactions. Randomly divide the data into training and testing sets in a 7:3 ratio, and construct the model through machine learning.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From date of randomization until the date of first documented date of death from anyh cause, whichever came first, assessed up to 100 months
  the time from the start of the trial until the patient died from all causes
Progression-free survival (PFS) | From date of randomization until the date of first documented progression, whichever came first, assessed up to 100 months
  From the time of trial initiation to the time of objective tumor progression or death.
Overall adverse event rate | up to 24 weeks
  According to the association evaluation of adverse drug reactions adopted by the National Adverse Drug Reaction Monitoring Center, the adverse drug reactions occurred in this study were classified into five levels: sure, probable, probable, suspicious and impossible.Adverse reactions with reference to the U.S. department of health and human services release of the common adverse reaction term evaluation criteria (CommonTerminologyCriteriaforAdverseEvents CTCAE) version 5.0
Incidence of grade III and above adverse events | up to 24 weeks
  According to the association evaluation of adverse drug reactions adopted by the National Adverse Drug Reaction Monitoring Center, the adverse drug reactions occurred in this study were classified into five levels: sure, probable, probable, suspicious and impossible.Adverse reactions with reference to the U.S. department of health and human services release of the common adverse reaction term evaluation criteria (CommonTerminologyCriteriaforAdverseEvents CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Yudong Qiu, Study Director — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School